CLINICAL TRIAL: NCT06604858
Title: Neoadjuvant Phase II Study of Pembrolizumab and Carboplatin Plus Paclitaxel for Stage I Triple-negative Breast Cancer (The TELESCOPE Study)
Brief Title: Neoadjuvant Pembrolizumab and Carboplatin Plus Paclitaxel for Stage I Triple-negative Breast Cancer
Acronym: TELESCOPE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MedSIR (Other)
Collaborators: Merk Sharp & Dohme España S.A. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MedOPP599; 2024-513511-27 (EudraCT Number)
Record Dates: First submitted 2024-09-17; First posted 2024-09-20 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Triple Negative Breast Cancer
Keywords: Breast Cancer; Stage I Triple Negative Breast Cancer; Pembrolizumab; Carboplatin; Paclitaxel
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — pembrolizumab; Carboplatin; Paclitaxel

STUDY DESIGN:
Intervention Model Description: Multicenter, single arm, non-comparative, phase II clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab and Carboplatin plus Paclitaxel (Experimental): Patients will receive treatment with Pembrolizumab and Carboplatin plus Paclitaxel up to surgery.
  The treatment is composed by 4 cycles of 21 days each (patients will be treated for a total of 84 days) and treatment will last until surgery.
  Interventions: Drug: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200 mg administered every three weeks intravenously on day 1 of each cycle.
Drug: Carboplatin — Carboplatin: area under the curve (AUC) 1.5, intravenously on day 1, day 8 and day 15 of each 21-days cycle.
Drug: Paclitaxel — Paclitaxel: 80 mg/m2, intravenously on day 1, day 8 and day 15 of each 21-days cycle.

SUMMARY:
This is a single arm, proof of concept phase II clinical trial to evaluate the combination of Pembrolizumab and Carboplatin plus Paclitaxel in patients with localized TNBC (tumor size ≥10 mm and up to 25 mm by mammogram and/or ultrasound, or ≤25 mm by breast MRI if performed within 2 weeks after biopsy, considering possible tissue inflammation post-procedure, as per local assessment), node-negative status (by clinical exam and local radiological evaluation) and who have not previously received chemotherapy, targeted therapy, and/or radiotherapy for invasive breast cancer.

DETAILED DESCRIPTION:
After signing informed consent form (ICF) and confirmed eligibility, eligible patients with localized TNBC, node-negative status, and who have not previously received chemotherapy, targeted therapy, and/or radiotherapy for invasive breast cancer (N=30) will receive treatment with Pembrolizumab and Carboplatin plus Paclitaxel up to surgery as indicated below:

* Pembrolizumab: 200 mg, every three weeks (Q3W), intravenously (IV) on day 1 (D1) of each cycle.
* Carboplatin: area under the curve (AUC) 1.5, IV on D1, D8 and D15 of each 21-days cycle.
* Paclitaxel: 80 mg/m2, IV on D1, D8 and D15 of each 21-days cycle.

The treatment is composed by 4 cycles of 21 days each (patients will be treated for a total of 84 days) and treatment will last until surgery.

Patients discontinuing the study treatment period will enter a post-treatment follow-up period during which survival and new anti-cancer therapy information will be collected, until end of study (EoS) or study termination, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent form (ICF) prior to beginning specific protocol procedures.
2. Female or male patients ≥ 18 years of age.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
4. Histologically confirmed TNBC as defined by the most ASCO/CAP guidelines based on local laboratory results.

   Note: TNBC means tumors that have <1 percent expression of Estrogen Receptor (ER) and Progesterone Receptor (PR) as determined by immunohistochemistry (IHC), and that are, for HER2, either 0 to 1+ by IHC, or IHC 2+ and fluorescence in situ hybridization (FISH) negative.
5. Node-negative status by clinical exam and local radiological evaluation.
6. Bilateral tumors and/or multi-focal (e.g, 2, separate lesions in the same quadrant)/multi-centric (e.g, 2 separate lesions in different quadrants) tumors are allowed. The tumor with the most advanced T stage should be used to assess the eligibility and TNBC needs to be confirmed for each breast/focus. In these cases, both axillae need to be assessed for nodal involvement confirmation.
7. No evidence of metastatic disease based on radiological assessment according to institutional practices.
8. No previous definitive ipsilateral breast surgery for the current breast cancer.
9. No prior chemotherapy, targeted therapy, and/or radiation therapy with therapeutic intent for this cancer.
10. Willingness to provide tumor tissue at baseline and at surgery and blood samples at the time of study entry (the closest time to the tumor biopsy), at C3D1, and at the end of treatment, prior to surgery (the closest time to the tumor biopsy).
11. Women of childbearing potential (WOCBP) must have a negative urine or serum pregnancy test and be willing to use an adequate method of contraception according to study protocol during treatment and for at least 4 months after the last dose of pembrolizumab. Female patients must refrain from egg cell donation and breastfeeding during treatment with pembrolizumab and for at least 4 months after the last dose of pembrolizumab.
12. Male patients and female patients of childbearing potential who engage in heterosexual intercourse must agree to use institution specified method(s) of contraception and must refrain from donating sperm or eggs during treatment with pembrolizumab and for at least 4 months after the last dose of pembrolizumab.
13. Patient has adequate bone marrow, liver, and renal function:

    * Hematological: White blood cell (WBC) count > 3.0 x 10 9/L, absolute neutrophil count (ANC) ≥ 1.5 x 10 9/L, platelet count ≥ 100.0 x10 9/L, and hemoglobin ≥ 9.0 g/dL (≥ 5.6 mmol/L).
    * Hepatic: total bilirubin ≤ institutional upper limit of normal (ULN) (except for Gilbert's syndrome); aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 times ULN.
    * Renal: serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
14. Patient must be accessible for treatment and follow-up.

Exclusion Criteria:

1. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
2. Has received prior systemic anti-breast cancer therapy, including an investigational agents or has used an investigational device within 4 weeks prior to allocation.
3. Has received prior taxane or platinum-based therapy.
4. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
5. Has had an allogenic tissue/solid organ transplant.
6. Has a history of invasive malignancy within the last 5 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer. For other cancers considered to have a low risk of recurrence, discussion with the Medical Monitor is required.
7. Participation in an interventional clinical study within 4 weeks of first dose of study treatment.
8. Major surgical procedure or significant traumatic injury within 14 days prior to enrolment or anticipation of need for major surgery within the course of the study treatment.
9. Has received a live vaccine within 30 days of first dose of study treatment.
10. Active autoimmune disease that has required systemic treatment in past 2 years, or ANY diagnosis of immunodeficiency or is receiving systemic steroid therapy (e.g, dosing exceeding 10 mg daily of prednisone or equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment. Replacement therapy (e.g, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
11. Current known infection with HIV, hepatitis B virus (HBV), or hepatitis C virus (HCV). Patients with past HBV infection or resolved HBV infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive hepatitis B core antibody [HBcAb] test, accompanied by a negative HBV DNA test) are eligible. Patients positive for HCV antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
12. Other active uncontrolled infection at the time of enrollment.
13. Significant cardiovascular disease within the last 6 months OR congestive heart failure (CHF) New York Heart Association (NYHA) Class II-IV or history of CHF NYHA Class III or IV.
14. History of (non-infectious) pneumonitis that required steroids or current pneumonitis.
15. Other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, contraindicate patient participation.
16. Pregnancy or breastfeeding or expecting to conceive children within the projected duration of the trial, starting with the screening visit through 6 months after the last dose of trial treatment.
17. Known hypersensitivity to the components of the study or its analogs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
To assess pathological complete response (pCR) rate in all patients. | From baseline up to 84 days (the date of breast surgery).
  To evaluate the pCR rate defined as the percentage of patients with ypT0/is, ypN0 at surgery based on local assessment.
  The efficacy will be evaluated by pCR rates concerning breast and lymph nodes (pCR breast + lymph node) in the overall population.

SECONDARY OUTCOMES:
To assess pathological complete response (pCR) rate according to PD-L1 status. | From baseline up to 84 days (the date of breast surgery).
  pCR rates will be calculated concerning breast and lymph nodes (pCR breast + lymph node) in patients with PD-L1 (+) tumors.
To evaluate residual cancer burden (RCB) at surgery. | At breast surgery.
  RCB score is a numeric index with numerical cutoffs to define the four classes (RCB-0: No carcinoma in breast or axillary lymph nodes; RCB-1; RCB-2; and RCB-3). RCB score will be calculated in the overall population at surgery.
To evaluate the incidence of adverse events [Safety and Tolerability]. | From baseline up to 84 days (the date of breast surgery).
  Incidence, severity, and relationship of treatment-emergent adverse events (TEAEs) based on local Investigator assessment as per NCI-CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Sara A Hurvitz, MD, Principal Investigator — Head of Hematology and Oncology Division, Fred Hutchinson Cancer Center, Seattle, WA (United States)
Locations (11):
- Spain (11):
  - Complejo Hospitalario Universitario A Coruña (CHUAC), A Coruña
  - Hospital Universitari Dexeus, Barcelona
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Institut Català d' Oncologia Girona (ICO), Girona
  - Hospital Universitario Clínico San Cecilio de Granada, Granada
  - Hospital Beata María Ana, Madrid
  - Hospital Cínico San Carlos, Madrid
  - Hospital Universitario de Navarra, Pamplona
  - Complejo Hospitalario Universitario de Santiago (CHUS), Santiago de Compostela
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Arnau de Vilanova de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Undecided